CLINICAL TRIAL: NCT06123156
Title: Intérêt de la rééducation érectile précoce Par Sildénafil après radiothérapie et Proctectomie Pour Cancer du Rectum : Essai contrôlé randomisé
Brief Title: Interest of Early Erectile Rehabilitation With Sildenafil After Radiotherapy and Proctectomy for Rectal Cancer
Acronym: RECTIL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/0398/HP; 2020-002682-34 (EudraCT Number)
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Sildénafil) (Active Comparator): Sildénafil during 10 months (50mg daily), start 30 days after surgery
  Interventions: Drug: Sildenafil
- Arm II (Placebo) (Placebo Comparator): Patients receive placebo during 10 month (1 platelet per day)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildénafil during 10 months (50mg daily), start 30 days after surgery
  Other Names: Arm I
  Arms: Arm I (Sildénafil)
Other: Placebo — 1 platelet during 10 months (daily), start 30 days after surgery
  Other Names: Arm II
  Arms: Arm II (Placebo)

SUMMARY:
This study aims to evaluate the efficacy of erectile rehabilitation with Sildenafil, in men treated with neoadjuvant proctectomy and radiotherapy for rectal cancer, in preventing long-term erectile dysfunction at 12 months post-operatively.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer in men in France, after lung and prostate cancer. Proctectomy (possibly preceded by radiotherapy) is the most effective treatment for this cancer, but erectile dysfunction (ED) is a frequent complication, even when the nerves are preserved during dissection, and has a major impact on the quality of life of operated men.

The cause of erectile dysfunction after rectal cancer surgery is usually neurological, due to intraoperative trauma to the autonomic nerves, while erectile dysfunction after radiotherapy is mainly vascular in origin, with damage to erectile tissue.

Several risk factors for sexual dysfunction after rectal cancer surgery have been reported (age, neoadjuvant radiotherapy, type of resection, operative difficulties and complications, body image affected by protective stoma). On the other hand, surgical expertise may be a protective factor.

In the physiological condition, the nitric oxide released by the pelvic nerves causes an increase in cyclic guanosine monophosphate, which in turn causes smooth muscle cells relaxation and an influx of blood into the cavernous body, triggering and maintaining the erection.

Similar to prostatectomy, nerve damage can occur during proctectomy through stretching, heat, ischemia or inflammation; this nerve damage results in reduced nitric oxide production.

Even in the absence of nerve damage, it has been demonstrated (in an animal model) that post-operative neurapraxia is responsible for the at least temporary disappearance of spontaneous and nocturnal erections, leading to cavernous hypoxia. This is followed by tissue changes (reduction in smooth and elastic muscle fibers in the corpora cavernosa, increase in collagen and endothelial dysfunction), which modify the hemodynamics of the carvernum body and ultimately lead to fibrosis of the erectile tissue.

These changes can become permanent despite subsequent nerve recovery, and are exacerbated by neoadjuvant radiotherapy. It is therefore important not to wait passively for erectile function to be restored, as lack of oxygenation to the corpora cavernosa can lead to permanent fibrosis and dysfunction.

This physiopathology is at the origin of the concept of erectile rehabilitation after prostatectomy, with the aim of maintain erections post-operatively and thus limiting fibrosis.

The benefits of erectile re-education after prostatectomy were first reported in 1997, with the early use of intracavernous injections of alprostadil. Following this study, various rehabilitation strategies have been recommended. Early treatment, i.e. within the first month, is recommended to promote cavernous oxygenation and prevent fibrosis.

The aims of rehabilitation are as follows :

* limit fibrosis;
* limit penis retraction and loss of height;
* oxygenate the cavernum body;
* preserve endothelial structure;
* preserve smooth muscle cell structure.

Various types of rehabilitation have been proposed: oral PDE-5 inhibitors, intra-cavernosal injections, urethral suppositories or vaccum.

PDE-5 inhibitors prevent the degradation of cyclic guanosine monophosphate, thus compensating for the reduction in nitric oxide and enabling a better erection.

Erectile rehabilitation using PDE-5 inhibitors could protect cavernous smooth muscle from irreversible pathophysiological changes. The basic concept is to administer a PDE-5 inhibitor at bedtime to facilitate nocturnal erections, which are thought to have a natural protective effect on the function of the cavernous bodies.

Padma-Nathan et al. reported the prospective administration of sildenafil 50 and 100 mg vs. placebo, daily and at bedtime, in patients undergoing nerve-sparing radical prostatectomy. After 36 weeks, erectile function was significantly better in the sildenafil group, with 27% responders, vs. 4% in the placebo group.

The mechanisms involved in erectile dysfunction after proctectomy for rectal cancer are similar to those of radical prostatectomy for prostate cancer.

The efficacy of PDE-5 inhibitors in the treatment of erectile dysfunction after proctectomy has already been demonstrated. However, its use as a preventive measure has rarely been reported.

Three studies have evaluated PDE-5 inhibitors in patients with erectile dysfunction after rectal resection, two of which used sildenafil (Viagra, Pfizer, New York, NY)

To our knowledge, only one study has evaluated the role of PDE-5 inhibitors (PDE-5i) in a preventive strategy.

Originality and innovation Despite the fact that sexual dysfunction is recognized as a frequent complication of rectal cancer treatment, there are currently no recommendations for its prevention and management.

In contrast to prostate cancer patients, information and treatment concerning erectile dysfunction (ED) are not systematically offered to men with colorectal cancer. The ability of sildenafil to facilitate the return of erections after radical prostatectomy has been demonstrated in several studies, and this treatment could benefit patients treated for rectal cancer.

To date, no randomized study has examined the usefulness of this early rehabilitation in patients managed for rectal cancer. This study proposes, for the first time, to evaluate the use of sildenafil after neo-adjuvant radiotherapy and surgery for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 70
* Patients undergoing surgery for cancer of the lower or middle rectum by total removal of the mesorectum with colorectal or coloanal anastomosis after neoadjuvant radiotherapy, with normal preoperative erectile function (defined by a combined IIEF erectile function domain score of at least 22).
* Nerve-conserving surgery
* Sexually active patient without treatment for erectile function prior to surgery
* Presence of a regular sexual partner (male or female)
* Adult having read and understood the information letter and signed the consent form
* Membership of a social security scheme

Exclusion Criteria:

* T4 tumor or tumor requiring extended surgery
* Patients with abnormal erectile function defined by a combined IIEF erectile function domain score of less than 22.
* History of prostate cancer
* Sleep disorders, patients taking sedatives/hypnotics
* Contraindication to SILDENAFIL EG 50 mg, film-coated tablet
* Contraindication to placebo
* Patients already treated with PDE5 inhibitors
* Patients suffering from SARS COV 2*
* Person deprived of liberty by an administrative or judicial decision or person placed under court protection / sub-guardianship or guardianship.
* Any history of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol, or to prevent the subject from giving informed consent.
* Person participating in another drug trial.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
the patient's response | 12 months postoperatively
  A patient is defined as a responder by a score of at least 22 for the erectile function domain of the International Index of Erectile Function (IIEF), comprising the six IIEF questions relating to erection (Q1-Q5 and Q15).

SECONDARY OUTCOMES:
IIEF erectile function domain score | Day 0, Month 1, Month 3, Month 6, Month 9, Month12
  Mesure of IIEF erectile function domain score, comprising the six IIEF erectile function questions (Q1-Q5 andQ15) at D0, M1, M3, M6, M9 and M12
International Index of Erectile Function (IIEF) global score | Day 0, Month 1, Month 3, Month 6, Month 9, Month 12
  International Index of Erectile Function (IIEF) global score measured at D0, M1, M3, M6, M9 and M12
Quality of life score | Day 0, Month 1, Month 3, Month 6, Month 9, Month 12
  Mesure of quality of life score (EORTC QLQ - C30 and QLQ - CR29) at D0, M1, M3, M6, M9 and M12
LARS score | Day 0, Month 1, Month 3, Month 6, Month 9, Month 12
  LARS score measured at D0, M1, M3, M6, M9 and M12
Fecal Continence Score | Day 0, Month 1, Month 3, Month 6, Month 9, Month 12
  Fecal Continence Score (Wexner score) measured at D0, M1, M3, M6, M9 and M12
Spontaneous erection evaluation | Month 1, Month 3, Month 6, Month 9, Month 12
  Number of patients with spontaneous erections on treatment at M3, M6, M9 and without treatment at M1, and M12
Benefits of psychological follow-up | after 10 months of treatment
  The number of patients with or without regular psychological follow-up. A patient is defined as having regular follow-up if he/she visits a psychologist and/or psychiatrist once or twice a month.
Compliance with treatment | after 10 months of treatment
  Number of unused tablets during the study. The patient will be considered as non-compliant if pill-taking over the entire 10-month treatment period is <80%.
Adverse and suspected adverse events | Month 1, Month 3, Month 6, Month 9, Month 12
  Number of AEs and SAEs in each group at M1, M3, M6, M9 and M12

IPD SHARING:
Plan to Share IPD: No